CLINICAL TRIAL: NCT06118944
Title: Visual Outcomes of a New Monofocal Intraocular Lens With Modified Optical Profile: a Randomized Controlled Clinical Study
Brief Title: Outcomes of Bilateral Implantation of an Enhanced Monofocal Intraocular Lens
Acronym: RCT_ICB00
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Trieste (Other)
Responsible Party: Principal Investigator, Daniele Tognetto, Professor, University of Trieste
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 202_2019
Record Dates: First submitted 2023-10-31; First posted 2023-11-07 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-10

CONDITIONS: Cataract
Keywords: IOL; intermediate distance; cataract surgery; enhanced monofocal
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- ICB00 Group (Experimental): ICB00 IOL
  Interventions: Device: ICB00 IOL
- ZCB00 Group (Active Comparator): ZCB00 IOL
  Interventions: Device: ZCB00 IOL
- CNA0T0 Group (Active Comparator): CNA0T0 IOL
  Interventions: Device: CNA0T0 IOL

INTERVENTIONS:
Device: ICB00 IOL — Bilateral implantation of ICB00 IOL
  Other Names: TECNIS EYHANCE IOL
  Arms: ICB00 Group
Device: ZCB00 IOL — Bilateral implantation of ZCB00 IOL
  Arms: ZCB00 Group
Device: CNA0T0 IOL — Bilateral implantation of CNA0T0 IOL
  Arms: CNA0T0 Group

SUMMARY:
To evaluate and compare the visual outcomes of an enhanced monofocal intraocular lens (IOL) with two different monofocal IOLs in patients scheduled for bilateral cataract surgery.

DETAILED DESCRIPTION:
The main objective of the study is the evaluation and comparison of the clinical outcomes of three parallel groups of patients after bilateral implantation of ICB00 IOL or ZCB00 IOL or CNA0T0 IOL respectively.

The ICB00 IOL is a modified monofocal IOL. Compared to other monofocal IOLs, its modified optical design was created to provide improved intermediate vision, comparable distance vision and a profile of dysphotopsia similar to other monofocal lenses.

Considering the modified optical profile of the ICB00 IOL, the primary objective will be the evaluation of visual performance at intermediate distance.

ELIGIBILITY:
Inclusion Criteria:

* clinically significant bilateral cataract (BCVA <20/40, cataract must be the primary cause of visual impairment)
* axial length between 21 and 27 mm
* the patient must be able to read, understand and provide written informed consent,
* the patient must be willing and able to comply with all study and follow-up procedures
* preoperative refractive cylinder ≤ 0.75 D

Exclusion Criteria:

* anterior segment pathology that could significantly affect results (e.g., chronic uveitis, iritis, corneal dystrophy, keratoconus)
* diabetic retinopathy
* uncontrolled glaucoma and/or intraocular pressure IOP> 24 mmHg
* all types of infections (acute eye disease, external/internal infection, systemic infection)
* traumatic cataract
* pupillary abnormalities including aniridia and/or pupil diameter in mesopic conditions in distance vision ≤ 2.5 mm and ≥ 6 mm
* microphthalmia
* amblyopia
* degenerative visual disorders (for example macular degeneration, optic nerve atrophy or retinal disorders)
* previous intraocular and corneal surgery
* systemic or ocular pharmacotherapy, which may impact visual acuity and/or cause floppy iris syndrome and/or insufficient dilation in the opinion of the investigator
* patients who are unable to fixate for a prolonged time (e.g. strabismus, nystagmus)
* period of pregnancy or breastfeeding for female patients

Ages: 50 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2019-11-11 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Bino DCIVA | 12 weeks after second eye surgery
  Binocular distance corrected intermediate visual acuity

SECONDARY OUTCOMES:
Mono DCIVA | 12 weeks after second eye surgery
  Monocular distance corrected intermediate visual acuity
Mono UIVA | 12 weeks after second eye surgery
  Monocular uncorrected intermediate visual acuity
Bino UIVA | 12 weeks after second eye surgery
  Binocular uncorrected intermediate visual acuity
Mono UDVA | 12 weeks after second eye surgery
  Monocular uncorrected distance visual acuity
Bino UDVA | 12 weeks after second eye surgery
  Binocular uncorrected distance visual acuity
Mono BCDVA | 12 weeks after second eye surgery
  Monocular best corrected distance visual acuity
Bino BCDVA | 12 weeks after second eye surgery
  Binocular best corrected distance visual acuity
Mono UNVA | 12 weeks after second eye surgery
  Monocular uncorrected near visual acuity
Bino UNVA | 12 weeks after second eye surgery
  Binocular uncorrected near visual acuity
Mono CNVA | 12 weeks after second eye surgery
  Monocular corrected near visual acuity
Bino CNVA | 12 weeks after second eye surgery
  Binocular corrected near visual acuity
Binocular defocus curves | 12 weeks after second eye surgery
  Binocular defocus curves in photopic conditions (from -4 D up to +2.00 D)
Catquest 9SF score changes | preop and 12 weeks after second eye surgery
  Changes in Catquest 9SF score before and 3 months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Daniele Tognetto, MD, Principal Investigator — University of Trieste
Locations (1):
- University Eye Clinic of Trieste, Trieste, Friuli Venezia Giulia, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lundstrom M, Behndig A, Kugelberg M, Montan P, Stenevi U, Pesudovs K. The outcome of cataract surgery measured with the Catquest-9SF. Acta Ophthalmol. 2011 Dec;89(8):718-23. doi: 10.1111/j.1755-3768.2009.01801.x. Epub 2009 Dec 21. PMID 20039853
- [Background] Ribeiro F, Cochener B, Kohnen T, Mencucci R, Katz G, Lundstrom M, Casanovas AS, Hewlett D. Definition and clinical relevance of the concept of functional vision in cataract surgery ESCRS Position Statement on Intermediate Vision: ESCRS Functional Vision Working Group. J Cataract Refract Surg. 2020 Feb;46 Suppl 1:S1-S3. doi: 10.1097/j.jcrs.0000000000000096. No abstract available. PMID 32126025